CLINICAL TRIAL: NCT05998863
Title: Effervescent Calcium Magnesium Citrate to Prevent Mineral Metabolism and Renal Complications of Chronic Proton Pump Inhibitor Therapy
Brief Title: EffCaMgCit to Prevent Mineral Metabolism and Renal Complications of Chronic PPI Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Khashayar Sakhaee, Professor, Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU-2023-0340
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Osteoporosis; Hypomagnesemia
Keywords: Bone mineral density
MeSH Terms: conditions — Osteoporosis | interventions — effervescent calcium magnesium citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To provide adequate blinding, each medication sachet will be labelled with the study name, IRB number, principal investigator's name, expiration date and identification number of the study subject. Labels will be applied to the appropriate medication sachets once the subject has been randomized and assigned to a treatment group. Labelling of the sachets will be done by personnel who are not engaged in patient care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EffCaMgCit (Experimental): 38 meq (760 mg) Ca, 20 meq (243 mg) Mg, and 100 meq total citrate per day; designed to be added to 6 oz water for 1-2 minutes, to be dissolved/suspended before swallowing.
  Interventions: Drug: EffCaMgCit
- Placebo (Placebo Comparator): Each sachet of Placebo will contain microcrystalline cellulose, but no calcium, magnesium or citrate. Placebo will be added to 6 oz water for 1-2 minutes, to be dissolved/suspended before swallowing.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: EffCaMgCit — Each sachet of EffCaMgCit will contain 19 meq or 380 mg calcium, 10 meq (122 mg) magnesium, and 50 meq total citrate.
  Other Names: Effervescent calcium magnesium citrate
  Arms: EffCaMgCit
Other: Placebo — Each sachet of Placebo will contain microcrystalline cellulose, but no calcium, magnesium or citrate.
  Arms: Placebo

SUMMARY:
Proton pump inhibitors (PPIs) are widely used for the control of gastric ulcer-gastritis, erosive esophagitis (gastroesophageal reflux disease), peptic ulcer disease (duodenal ulcer), and heartburn. Despite their efficacy, their use has been implicated in possibly causing fragility fractures (osteoporosis), hypomagnesemia (magnesium deficiency) and increased risk of chronic kidney disease (CKD). The current trial represents the investigators ongoing effort to discern whether these complications could be averted by effervescent calcium magnesium citrate (EffCaMgCit).

DETAILED DESCRIPTION:
In the current proposal, the investigators wish to conduct a 1-year treatment trial, directed at obtaining more definitive evidence that EffCaMgCit overcomes all three complications of PPI.

Aim 1. To test the hypothesis that EffCaMgCit would prevent/treat osteoporosis, by suppressing parathyroid function and bone resorption, thereby stabilizing bone mineral density (BMD). The critical endpoint will be overall change in BMD T-Score and Z-Score from baseline to the end of study. Secondary endpoints will be the change in serum PTH and C-terminal telopeptide (CTX).

Aim 2. To test the hypothesis that EffCaMgCit would prevent/treat hypomagnesemia/magnesium deficiency, by providing bioavailable magnesium. The critical endpoint will be the overall change in the fractional excretion of magnesium (FEMg) and free muscle magnesium by MRS from baseline to the end of study. Secondary endpoints will be the change in serum and urinary magnesium.

Aim 3. To test the hypothesis that EffCaMgCit would reduce the risk of CKD during PPI use by averting putative hypomagnesemia/magnesium deficiency and neutralizing acid load. The investigators propose that PPI causes hypomagnesemia/magnesium deficiency and confers an acid load, - factors implicated for incident CKD and its progression. EffCaMgCit is expected to avert incident CKD by providing bioavailable magnesium and alkali load. Critical endpoints will be the overall change in endogenous creatinine clearance, urinary alpha-1 microglobulin, and a measure of acid-base status.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory adult subjects (> 21 years of age) of either gender of any ethnicity
* Must have taken PPI (omeprazole or equivalent ≥ 20 mg/day, ≥ three times per week, for at least 2 months)
* Expected to continue at a similar dosage
* Stage 1 hypertension (with systolic blood pressure <140 and diastolic <90)
* Controlled diabetes mellitus Type II with HbA1C less than 7%

Exclusion Criteria:

* End-stage renal failure on dialysis
* Hypercalcemia,
* Hypophosphatemia (serum P < 2.5 mg/dL)
* Hypertension stage 2 or higher
* Diabetes Type II with HbA1C ≥ 7%
* Treatment with adrenocorticosteroids, diuretics, non-steroidal anti-inflammatory agents - - Regular dose of magnesium supplements, bisphosphonate, teriparatide, denosumab or selective estrogen receptor modulators
* Required to take calcium

Inclusion/exclusion of other drugs or conditions will be considered on an individual basis.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Bone Mineral Density (BMD) T-Score at 1 Year | Baseline and 1 year
  Change in Bone Mineral Density (BMD) T-Score from baseline to 1 Year as measured by dual photon absorptiometry. The range, as defined by the World Health Organization (WHO), for T-Score is: -1 and above = Normal, Between -1 and -2.5 = Osteopenia, -2.5 and below = osteoporosis.
Change From Baseline in the Fractional Excretion of Magnesium (FEMg) at 1 Year | Baseline and 1 year
  Change From Baseline in the Fractional Excretion of Magnesium (FEMg) at 1 Year as measured by the ratio of magnesium clearance and creatinine clearance, using 24-h urinary magnesium and creatinine and corresponding serum magnesium and creatinine obtained post meal/load.
Change from baseline in endogenous creatinine clearance at 1 year. | Baseline and 1 year
  Change from baseline in endogenous creatinine clearance at 1 year. Endogenous creatinine clearance will be obtained by using 24-h urinary creatinine and post-meal/load venous blood sample ((uCr, mg/24hr) / (sCr, mg/dL * 14.4)) as well as using the Cockcroft and Gault formula ([(140 - age) x TBW] / (Scr x 72) (x 0.85 for females)).
Change From Baseline in Bone Mineral Density (BMD) Z-Score at 1 Year | Baseline and 1 year
  Change From Baseline in Bone Mineral Density (BMD) Z-Score at 1 Year as measured by dual photon absorptiometry. Outcome is considered positive if the Z Score after one year of treatment becomes less negative (less than -2). There is no specific score range for the Z Score.
Change From Baseline in Free Muscle Magnesium at 1 Year | Baseline and 1 year
  Change From baseline in free muscle magnesium at 1 year as assessed by measuring intracellular Mg in a calf muscle, by using 31P (Phosphorous) magnetic resonance spectroscopy (MRS).

SECONDARY OUTCOMES:
Change in Serum Parathyroid Function (PTH) | Baseline and 1 year
  Change from baseline in serum parathyroid function (PTH) at 1 year will be measured by Biomerica Intact-PTH ELISA.
Change in C-terminal telopeptide (CTX) | Baseline and 1 year
  Change from baseline in serum bone resorption marker C-terminal telopeptide (CTX) at 1 year will be measured by lab finding utilizing ELISA CTX-I (CrossLaps).
Change in Serum Magnesium | Baseline and 1 year
  Change from baseline in serum magnesium at 1 year will be measured by ion selective electrode.
Change in Urine Magnesium | Baseline and 1 year
  Change from baseline in urine magnesium at 1 year measured by atomic absorption.

CONTACTS AND LOCATIONS:
Overall Officials: Khashayar Sakhaee, MD, Principal Investigator — UTSW
Locations (2):
- United States (2):
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No